CLINICAL TRIAL: NCT07041983
Title: Effects of Anti-obesity Medications on 24h Energy Metabolism and Body Composition in Patients With Obesity
Brief Title: 24-h Energy Expenditure and Anti-obesity Medication
Acronym: SEM-TIR
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Alessio Basolo, Researcher, University of Pisa
Other Study IDs: SEM-TIR; 539901_2019_Santini_PRIN2017 (Other Grant/Funding Number: Italian Ministry of the University)
Record Dates: First submitted 2025-05-28; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Obesity
Keywords: energy metabolism; body composition
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- antiobesity medication and energy expenditure: patients with obesity for the administration anti-obesity medication (Semaglutide or Tirzepatide) for the clinical use.
  Interventions: Drug: anti obesity medication

INTERVENTIONS:
Drug: anti obesity medication — Patients with obesity or overweight, with at least one weight-related comorbidity who are expected to start treatment with Semaglutide (Wegovy) or Terzepatide (Mounjaro) at enrolment will be eligible to enrol into the study.
  Patients will be treated and observed according to normal clinical practice. Participation in this study does not limit the physicians' clinical decision making as to the most appropriate treatment for the patient during the course of the study

SUMMARY:
This study investigates the long-term effects of anti-obesity medications (Semaglutide and Tirzepatide) on energy metabolism (24-hour energy expenditure and substrate oxidation) and body composition via Dual-energy X-ray absorptiometry (DXA)

DETAILED DESCRIPTION:
This study will explore the long-term effects of obesity treatments, including anti-obesity medications (AOMs) such as GLP-1 receptor agonist (Semaglutide) and GIP/GLP-1 receptor agonist (Tirzepatide), on energy metabolism (24-hour energy expenditure and substrate oxidation), body composition (fat mass and fat-free mass). The study will include AOMs may lead to a state of metabolic adaptation, one of the reasons for weight regain. To date, no studies have assessed the effects of AOMs on 24-hour energy expenditure measured by using the metabolic chamber.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >= 30 kg/m² or >= 27 kg/m² with at least one weight-related comorbidity and stable body weight (±2 kg in prior 3 months)
* informed consent, adherence to study protocol, negative pregnancy test and contraception use (if applicable), and absence of cardiovascular events or end-organ damage.

Exclusion Criteria:

* psychiatric conditions impairing adherence, history of medullary thyroid cancer, pregnancy/lactation
* diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-75 years with Body mass index (BMI) >= 30 kg/m² or >= 27 kg/m² with at least one weight-related comorbidity (e.g., prediabetes, hypertension, dyslipidemia, sleep apnea, cardiovascular disease) and stable body weight (±2 kg in prior 3 months)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
change in 24h energy expenditure after 6 months of treatment | Baseline and 6 months after treatment initiation
  measurement of 24-hour energy expenditure (kilocalories) by using the metabolic chamber (whole room indirect calorimeter) at baseline and after 6 months of treatment

SECONDARY OUTCOMES:
Change in body composition | Baseline and 6 months after treatment initiation
  Quantification of variations in fat mass and fat-free mass (kg) following 6 months of therapy, as determined by Dual-Energy X-ray Absorptiometry (DEXA)